CLINICAL TRIAL: NCT06437470
Title: Combined Effect Of Blood Flow Restriction Technique And Conventional Physical Therapy Program After Anterior Cruciate Ligament Reconstruction
Brief Title: Effect of Blood Flow Restriction Technique After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Ali Abed, Assistant Lecturer of Physical Therapy for Musculoskeletal System Disorders and its Surgery, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005176
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A triple-blinded randomized controlled trial will be conducted, ensuring that participants, the research assistant (who serves as the examiner for all participants) and the statistician are blinded to the treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy program (Sham Comparator): participants will receive the conventional physical therapy program while using non-inflated cuff as a sham treatment during exercising.
  Interventions: Other: blood flow restriction technique
- blood flow restriction combined to conventional physical therapy program (Experimental): participants will receive the conventional physical therapy program with the use of BFR cuff which will be inflated to reach 80% of limb occlusive pressure
  Interventions: Other: blood flow restriction technique

INTERVENTIONS:
Other: blood flow restriction technique — All participants in the control group will receive the conventional physical therapy program with the use non-inflated cuff as a sham treatment during exercising.
  All participants in the intervention group will receive the conventional physical therapy program combined to blood flow restriction to 80% of limb occlusive pressure by using blood flow restriction cuff.

SUMMARY:
The purpose of this study will be to evaluate the effect of adding BFR (using 80% of LOP) to the conventional physical therapy program on knee function, functional test, balance, quadriceps and hamstrings muscles strength, thigh muscle girth and knee effusion in rehabilitation after ACLR.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury is one of the most common knee injuries especially in the age range 20 to 29 years. It is commonly seen during sport activities including jumping, pivoting or during contact with the other players (Khalil et al., 2023).

Quadriceps and hamstrings muscle weakness and atrophy are commonly seen after Anterior cruciate ligament reconstruction (ACLR) mainly due to weight bearing limitation in the early stage of rehabilitation (Barber-Westin and Noyes 2019 and Hughes et al., 2019). Recent rehabilitation protocols focused on range of motion (ROM) exercises and increased muscle activation in the early post-operative phase to minimize complications such as joint stiffness and muscle weakness (Myer et al., 2006 and Patterson et al., 2019a).

It is recommended by the American College of Sports Medicine to use 60% to 70% of one repetition maximum (1 RM) to increase muscle strength and 70% to 80% of 1 RM to increase muscle size. However, using these percentage of loads in the early post-operative phase after ACLR may not be applicable (Barber-Westin and Noyes 2019). Therefore, therapists considered it is necessary to find a safe exercise protocol designed to increase muscle strength and mass to be used in the early post-operative phase. One of these protocols is the blood flow restriction training (BFRT) (Patterson et al., 2019a).

The BFRT is a technique that restricts arterial and venous circulation in the working muscles during exercise (Scott et al., 2015). This technique uses a pneumatic tourniquet system that applies external pressure to the most proximal part of the arm or the thigh. Cuff inflation causes compression on the vascular structures under the cuff leading to occlusion of the venous return and restriction of the arterial blood flow to the distal part of the limb. This intentionally induced ischemic environment results in a state of hypoxia within the distal muscles (Manini and Clark 2009). In such environment, muscle strength and hypertrophy can be reached by smaller external loads such as 20% or 30% of 1RM (Loenneke et al., 2012a). This makes the BFRT applicable in the early post-operative phase of rehabilitation without stressing the knee joint, thus protecting the graft and minimizing the risk of increasing any associated injuries in cartilage or meniscus (Loenneke et al., 2012b and Arve et al., 2020).

The BFRT is beneficial for many groups such as geriatrics and those with degenerative joint diseases, ligamentous injury and inflammatory diseases (Hughes et al., 2017). Early BFRT research designs used general measures to calculate cuff pressures, such as setting pressure relative to systolic blood pressure, thigh circumference, or random pressures which is probably inaccurate especially with change in limb circumference or body position (Takano et al., 2005 and Loenneke et al., 2015). A study performed by (Khalil et al., 2023) used the portable doppler ultrasound device to calculate limb occlusion pressure (LOP) of dorsalis pedis artery while manually inflating the restriction cuff. This procedure is operator dependent and may lead to some errors, especially in determining the exact location of the artery.

Recent research recommends the use of individualized BFRT where the percentage of occlusion of the vascular structures is determined automatically for each individual separately (Scott et al., 2015).

Previous studies concluded that BFRT after ACLR was effective in improving knee extension and flexion torques, pain, and balance (Spada et al., 2022, Bobes et al., 2020 and Jung et al., 2022) A recent systematic review performed by (Colapietro et al., 2023) found that limited studies included functional testing of the knee joint after BFRT which will be covered in this study using the latest wireless version of AirBands produced by VALD performance company which possesses the ability to automatically calculate LOP for each participant alone as recommended by the guidelines of Australian Institute of Sport.

Up to the authors' knowledge, there was no study has investigated the effect of blood flow restriction (BFR) using 80% of LOP combined with the conventional physical therapy program on knee function and balance compared to the conventional physical therapy program alone after ACLR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18-35 years.
2. Underwent an ACLR semitendinosus autograft one-week post-operative
3. Willingness to participate in the intervention and subsequent assessment.
4. BMI from 18.5 to 29.9 kg/m2.

Exclusion Criteria:

1. Insecure graft fixation (due to bone quality, suspension).
2. Active infection.
3. Postsurgical excess knee swelling that may limit exercise performance.
4. ACLR using bone tendon bone (BTB) graft.
5. Any cardiovascular disease such as hypertension.
6. Any lower limb trauma.
7. Hip and ankle pathology.
8. BMI more than 30 kg/m2

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
knee function | after 3 months of intervention
  will be assessed by the Arabic version of the knee outcome survey-activities for daily living scale.
  It encompasses six questions addressing restrictions in daily activities caused by symptoms like pain, swelling, and instability, and eight questions evaluating difficulties in functional tasks such as walking, stair climbing, and sitting or standing up from a chair.
  Each question is rated on a 6-point Likert scale.
  Scores range from 0 to 70, with higher scores indicating better functional capacity.
knee functional test | after 3 months of intervention
  will be assessed by the single leg hop test
balance | after 3 months of intervention
  will be assessed by the Y balance test for the lower quarter
quadriceps and hamstring muscles strength | after 3 months of intervention
  will be assessed by the hand held dynamometer

SECONDARY OUTCOMES:
Thigh muscle girth | baseline then 3 months after intervention
  will be assessed by a non-elastic measuring tape
Knee effusion | baseline then 3 months after intervention
  will be assessed by a non-elastic measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Enas F Youssef, Professor, Study Chair — Prof. of PT for Musculoskeletal System Disorders and its Surgery, Faculty of PT, Cairo University; Dina S Abd Allah, lecturer, Study Director — Lec. of PT for Musculoskeletal System Disorders and its Surgery, Faculty of PT, Cairo University; Ahmed S Elkalyoby, Asst. prof, Study Director — Asst. prof. of orthopedic surgery, Cairo University
Locations (1):
- Faculty of physical therapy - Cairo University, Cairo, Giza Governorate, Egypt